CLINICAL TRIAL: NCT06147375
Title: Efficacy and Safety of Immunosuppressive Withdrawal After Pediatric Liver Transplantation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wei Gao (Other)
Responsible Party: Sponsor-Investigator, Wei Gao, Head of Department of Pediatric Organ Transplantation, Tianjin First Central Hospital
Organization: Tianjin First Central Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023DZX32
Record Dates: First submitted 2023-10-26; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Immune Tolerance; Immunosuppression; Liver Transplant; Complications
Keywords: Immune Tolerance; Pediatric liver transplant; Immunosuppression
MeSH Terms: interventions — Tacrolimus; Cyclosporine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- immunosuppressive withdrawal (Experimental): After enrollment,the recipients will take IS withdrawal follow the protocol of this study.Following enrollment, recipients will be examined at several time periods such as peripheral blood test,liver function , liver biopsy, and other relevant indicators to determine immunosuppressant withdrawal condition and adverse effects.
  Interventions: Drug: Tacrolimus or Cyclosporine A

INTERVENTIONS:
Drug: Tacrolimus or Cyclosporine A — The protocol of IS withdrawal:Week 1-4 take Tacrolimus (Tac) or Cyclosporine A (CsA) once daily for weeks. Week 5-8 medication reduction to taking Tac / CsA 4 times a week . Week 9-12 reduction to taking Tac/ CsA 3 times a week. Week 13-18 reduction to taking Tac / CsA 2 times a week . Week 19-24 reduction to taking Tac/ CsA once per week. Week 25, the recipients will stop taking Tac/ CsA.
  Other Names: immunosuppression withdrawal

SUMMARY:
The goal of this clinical trial is to learn about the efficacy and safety of immunosuppressive withdrawal in pediatric liver transplant recipients. The main question it aims to answer is:exploring the landscape of immune tolerance after pediatric liver transplantation. Moreover,this clinical trial aims to provide important foundation and clinical data for inducing immune tolerance, as well as to clarify the mechanism of immune tolerance development in pediatric liver transplantation, identify biomarkers that can be used to predict immune tolerance, and build a prediction model of immune tolerance after pediatric liver transplantation.

The study planned to enroll 47 recipients after pediatric liver transplantation which would gradually withdrawal immunosuppressive after enrollment, divided the participants into immune tolerance and immune intolerance groups based on the outcome of immunosuppressive withdrawal.In this study, we collect the peripheral blood and liver biopsy samples from the two groups, find biomarkers with predictive value for immune tolerance in recipients after pediatric liver transplantation, and build a predictive model of immune tolerance by machine learning.

DETAILED DESCRIPTION:
Background: The main conditions which require pediatric liver transplantation are benign diseases with curable primary diseases, such as metabolic and biliary diseases. After liver transplantation, the two main risk factors affecting recipients survival are cumulative IS toxicity and chronic graft injuries. Adverse reactions such as renal dysfunction, metabolic problems, infection, and cancer can result from chronic exposure to IS. As a result, decreasing or stopping immunosuppressive treatment is an effective way for improving recipients survival after liver transplantation. Currently, the recipients after pediatric liver transplantation lacks defined IS withdrawal plans and also unified and uniform recipients selection criteria and processes. Additionally, IS withdrawal could result in graft fibrosis, rejection, and graft dysfunction.Therefore, the safety and efficacy of IS withdrawal needs to be discussed.

Methods:The study planned to enroll 47 recipients after pediatric liver transplantation which would gradually withdrawal IS after enrollment, divided the participants into immune tolerance and immune intolerance groups based on the outcome of IS withdrawal.In this study, we will collect the peripheral blood and liver biopsy samples from the two groups, find biomarkers with predictive value for immune tolerance in recipients after pediatric liver transplantation, and build a predictive model of immune tolerance by machine learning.

Protocol after enrollment: After enrollment,the recipients will take IS withdrawal follow the protocol of this study.The IS withdrawal protocol is once daily for weeks 1 to 4, then decreased every 4 weeks until the IS is totally stopped by 25 weeks. Following enrollment, recipients will be examined at several time periods such as peripheral blood tests,liver function , liver biopsy, and other relevant indicators to determine IS withdrawal and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Age at liver transplantation: under 6 years
* Follow-up time after liver transplantation: more than 4 years
* Liver function maintains normal before enrollment
* Monotherapy of IS (Tacrolimus or Cyclosporine A)
* Liver biopsy: No signs of acute rejection or chronic rejection, and no obvious fibrosis (Ishak<2) 2 years before enrollment
* Female recipients of fertility treatment must have a negative pregnancy test before enrollment
* No Hepatitis virus infection 1 year before enrollment
* Written consents are required

Exclusion Criteria:

* Original disease before liver transplantation: Tumor, secondary liver transplantation, hepatitis virus infection, autoimmune hepatitis
* Type of liver transplantation: ABO incompatible liver transplantation or multiple organ transplantation
* Liver biopsy: obvious fibrosis(Ishak≥2；LAFSc moderate or severe)
* Recipients taking IS for other diseases besides their liver transplantation

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of immune tolerance participants | Enrollment to 2 year post cessation of immunosuppression
  Number of participants who are immune tolerance, defined as those who successfully withdraw from immunosuppression and maintain normal graft status as assessed by liver biopsy and liver tests 2 years after complete immunosuppression withdrawal.

SECONDARY OUTCOMES:
Number of participants with complications attributed to immunosuppression withdrawal | Enrollment to 4 year post cessation of immunosuppression
  This endpoint is comprised of complications related to immunosuppression withdrawal and is defined as the occurrence of any of the following: death or graft loss, histologic evidence of refractory acute rejection or biopsy confirmed chronic rejection.
Impact of iImmunosuppression withdrawal on graft histology | Enrollment to 4 year post cessation of immunosuppression
  Histologic progression determined from the stage of fibrosis at baseline to completion of the study according to the Ishak Severity System
Severity of acute rejection in immunotolerant recipients | Enrollment to 2 year post cessation of immunosuppression
  Acute rejection severity (mild, moderate, severe) is based on the Banff global assessment grade according to the central pathology reading of the liver biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Gao, MD, Principal Investigator — Tianjin First Central Hospital
Locations (1):
- Tianjin First Central Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No